CLINICAL TRIAL: NCT03948763
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety and Tolerability of mRNA-5671/V941 as a Monotherapy and in Combination With Pembrolizumab in Participants With KRAS Mutant Advanced or Metastatic Non-Small Cell Lung Cancer, Colorectal Cancer or Pancreatic Adenocarcinoma
Brief Title: A Study of mRNA-5671/V941 as Monotherapy and in Combination With Pembrolizumab (V941-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V941-001; V941-001 (Other: MSD Protocol Number)
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms
Keywords: cancer; solid tumors; therapeutic vaccine; Pembrolizumab; PD1; PD-1; PDL1; PD-L1; KRAS; mRNA
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: V941 Monotherapy (Experimental): V941(mRNA-5671/V941) 1 mg administered intramuscularly (IM) once every 3 weeks (Q3W) for 9 3-week cycles
  Interventions: Biological: V941
- Part 1: V941 + Pembrolizumab (Experimental): V941(mRNA-5671/V941) 1 mg administered IM Q3W for 9 3-week cycles and pembrolizumab 200 mg, intravenous (IV) for 35 3-week cycles
  Interventions: Biological: V941; Biological: Pembrolizumab
- Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) (Experimental): V941(mRNA-5671/V941) 1 mg administered IM Q3W for 9 3-week cycles and pembrolizumab 200 mg, IV for 35 3-week cycles
  Interventions: Biological: V941; Biological: Pembrolizumab
- Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) (Experimental): V941(mRNA-5671/V941) 1 mg administered IM Q3W for 9 3-week cycles and pembrolizumab 200 mg, IV for 35 3-week cycles
  Interventions: Biological: V941; Biological: Pembrolizumab
- Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab) (Experimental): V941(mRNA-5671/V941) 1 mg administered IM Q3W for 9 3-week cycles and pembrolizumab 200 mg, IV for 35 3-week cycles
  Interventions: Biological: V941; Biological: Pembrolizumab

INTERVENTIONS:
Biological: V941 — V941 administered IM, Q3W for 9 3-week cycles
  Other Names: mRNA-5671/V941
Biological: Pembrolizumab — Pembrolizumab 200 mg, IV for 35 3-week cycles
  Other Names: MK-3475
  Arms: Part 1: V941 + Pembrolizumab; Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab); Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab); Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)

SUMMARY:
This study will determine the safety and tolerability and establish a preliminary recommended Phase 2 dose of V941(mRNA-5671/V941) as a monotherapy and in combination with pembrolizumab infusion.

ELIGIBILITY:
Inclusion Criteria:

Part 2 Only

- Has a histologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC), non-mismatch repair deficient/microsatellite instability-high tumors colorectal cancers (non-MSI-H CRC), or pancreatic adenocarcinoma, and confirmed HLA types HLA-A11:01 and/or HLA C08:02 (and/or potentially other additional HLA types to be specified).

NSCLC: Participants must have been tested for mutations affecting EGFR and/or anaplastic lymphoma kinase (ALK). Participants with ALK or epidermal growth factor receptor (EGFR)-positive NSCLC must have had recurrent or progressive disease (PD) after treatment with the corresponding inhibitor and current standard of care, in any sequence.

Non-MSI-H CRC: Participant tumors must have been locally tested for MSI and have been found to be non-MSI-H.

All

* Has a histologically confirmed advanced or metastatic KRAS 4MUT+ (G12D, G12V, G13D or G12C) (4 prevalent KRAS mutant antigens in solid tumors) solid tumor identified by local laboratory testing, and who have received, or been intolerant to, or ineligible for all treatment known to confer clinical benefit.
* A male participant must agree to use study-approved contraception during the treatment period and for at least 120 days after the last dose of study intervention and refrain from donating sperm during this period.
* A female participant was not be pregnant, not breastfeeding, and at not be a woman of childbearing potential (WOCBP) OR if a WOCBP, agrees to follow study-approved contraceptive guidance during treatment period and for at least 120 days after the last dose of study intervention.
* Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* For Part 1 only: Cutaneous lesions can be considered in addition to imaging, but measurable disease should be defined by radiologic assessment.
* Have an evaluable archival tumor sample to submit for analysis. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
* Have adequate organ function
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization or treatment allocation
* Has an active infection requiring therapy.
* Has a history of interstitial lung disease.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy.
* Has not fully recovered from any effects of major surgery or has evidence of detectable infection. Surgeries that required general anesthesia must be completed at least 2 weeks before first study treatment administration. Surgery requiring regional/epidural anesthesia must be completed at least 72 hours before first study treatment administration and participants should be recovered.
* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study therapy, non-cytotoxic small molecule therapeutics within 5 half-lives (or 2 weeks, whichever is longer) prior to the first dose of study treatment, or has not recovered to Common Toxicity Criteria for Adverse Events (CTCAE) Grade 1 or better from any adverse events that were due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related adverse events).
* Has received a live-virus vaccine within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Has received hematopoietic colony-stimulating growth factors (eg, granulocyte-colony stimulating factor, granulocyte-macrophage-colony stimulating factor, macrophage colony stimulating factor) within 2 weeks prior to the first dose of study intervention.
* Discontinued from therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (TCR; eg, cytotoxic T lymphocyte-associated antigen 4 (CTLA-4), CD137 (4-1BB, Tumor necrosis factor-receptor superfamily 9 [TNFSF9]), and OX 40 (TNFRSF4), due to a Grade 3 or higher immune-related adverse event (irAE).
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 28 days prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection.
* Has a known history of HIV.
* Has a known psychiatric or substance abuse disorder that would interfere with cooperating with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (26):
- United States (10):
  - Banner MD Anderson Cancer Center ( Site 1008), Gilbert, Arizona
  - City of Hope ( Site 1002), Duarte, California
  - University of California at San Francisco ( Site 1006), San Francisco, California
  - Smilow Cancer Hospital at Yale New Haven ( Site 1005), New Haven, Connecticut
  - Dana-Farber Cancer Institute (Boston) ( Site 1007), Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada ( Site 1012), Las Vegas, Nevada
  - Tennessee Oncology Nashville Drug Development Unit ( Site 7000), Nashville, Tennessee
  - START San Antonio ( Site 1004), San Antonio, Texas
  - Baylor Scott & White Medical Center - Temple ( Site 1009), Temple, Texas
  - Northwest Medical Specialties, PLLC ( Site 1001), Tacoma, Washington
- Australia (3):
  - Kinghorn Cancer Centre ( Site 6000), Darlinghurst, New South Wales
  - Southern Oncology Clinical Research Unit SOCRU ( Site 6002), Bedford Park, South Australia
  - Monash Health-Monash Medical Centre ( Site 6001), Clayton, Victoria
- Hong Kong (2):
  - Prince of Wales Hospital ( Site 2002), Hong Kong
  - Queen Mary Hospital ( Site 2001), Hong Kong
- New Zealand (2):
  - New Zealand Clinical Research (Christchurch) ( Site 6501), Christchurch, Canterbury
  - Auckland City Hospital ( Site 6500), Auckland
- Singapore (3):
  - National University Hospital ( Site 3006), Singapore, Central Singapore
  - National Cancer Centre Singapore ( Site 3005), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 3007), Singapore, Central Singapore
- South Korea (3):
  - Asan Medical Center ( Site 0802), Songpagu, Seoul
  - Seoul National University Hospital ( Site 0801), Seoul
  - Severance Hospital ( Site 0800), Seoul
- Taiwan (3):
  - National Cheng Kung University Hospital ( Site 4002), Tainan
  - National Taiwan University Hospital ( Site 4000), Taipei
  - Taipei Veterans General Hospital ( Site 4001), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Started | 3 | 15 | 20 | 16 | 16
Participants Switched Over From V941 Monotherapy to V941 + Pembrolizumab | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 15 | 20 | 16 | 16
Not completed — Sponsor's decision | 0 | 2 | 6 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Death | 2 | 12 | 13 | 10 | 11
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab) | Total
Number analyzed (Participants) | 3 | 15 | 20 | 16 | 16 | 70
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 2 | 10 | 9 | 12 | 6 | 39
  >= 65 years | 1 | 5 | 11 | 4 | 10 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 13 | 7 | 9 | 39
  Male | 2 | 6 | 7 | 9 | 7 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 3 | 11 | 19 | 15 | 16 | 64
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 12 | 9 | 9 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2
  White | 2 | 12 | 8 | 6 | 7 | 35
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS where ECOG PS Grade 0 is fully active, able to carry on all pre-disease performance without restriction. Grade 1 is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    ECOG = 0 | 2 | 7 | 1 | 7 | 6 | 23
    ECOG = 1 | 1 | 8 | 19 | 9 | 10 | 47
Primary Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma of the Colon | 0 | 1 | 0 | 0 | 0 | 1
  Adenocarcinoma of the Pancreas | 0 | 1 | 0 | 0 | 6 | 7
  Carcinoma Of Ampulla of Vater | 0 | 1 | 0 | 0 | 0 | 1
  Cholangiocarcinoma | 0 | 1 | 0 | 0 | 0 | 1
  Colorectal Cancer, not otherwise specified | 2 | 7 | 0 | 16 | 0 | 25
  Lung Cancer, not otherwise specified | 1 | 0 | 0 | 0 | 0 | 1
  Pancreatic Cancer (Not Islets) | 0 | 3 | 0 | 0 | 10 | 13
  Rectal | 0 | 1 | 0 | 0 | 0 | 1
  Non-Small Cell Lung Cancer, not otherwise specified | 0 | 0 | 20 | 0 | 0 | 20
Prior Line of Therapy [Count of Participants; unit: Participants]
  First Line | 1 | 2 | 5 | 0 | 1 | 9
  Second Line | 2 | 5 | 5 | 4 | 5 | 21
  Third Line | 0 | 2 | 5 | 6 | 7 | 20
  Fourth Line | 0 | 3 | 1 | 2 | 3 | 9
  Fifth Line or Greater | 0 | 3 | 4 | 4 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Dose-Limiting Toxicities (DLTs)
Description: The following toxicities graded for severity using National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE), were considered a DLT if judged by the investigator to be possibly related to study investigational products: 1) Grade 4 nonhematologic toxicity (ie. not a laboratory finding). 2) Grade 4 hematologic toxicity lasting ≥ 7 days, except thrombocytopenia: 3) Grade 4 thrombocytopenia of any duration 4) Grade 3 thrombocytopenia associated with clinically significant bleeding 5) Any nonhematologic AE ≥ Grade 3 in severity, with some exceptions 6) Any Grade 3 or Grade 4 nonhematologic laboratory value that meets one of the study criteria 7) Febrile neutropenia Grade 3 or Grade 4 8) Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity. 9) Any treatment-related toxicity that causes participant to discontinue treatment during Cycle 1. 10) Grade 5 toxicity 11) Any other clinically significant toxicity judged to be a DLT by investigator.
Time Frame: Cycle 1 (Up to 21 days)
Population: The DLT evaluable population included all participants who received at least 1 dose of study treatment and were either observed for safety for 21 days after the first dose of treatment or experienced a DLT prior to 21 days after the first dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 2 | 14 | 0 | 0 | 0
Participants | 0 | 0 |  |  |

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 27 months
Population: All participants who received at least 1 dose of study treatment. For AEs which occurred during Part 1 prior to switch-over, the information is in the Part 1: V941 Monotherapy column. For AEs which occurred during Part 1 subsequent to switch-over, the information is in the Part 1: V941 + Pembrolizumab column.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 3 | 16 | 20 | 16 | 16
Participants | 3 | 15 | 20 | 16 | 16

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to approximately 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 3 | 16 | 20 | 16 | 16
Participants | 0 | 1 | 1 | 2 | 3

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experienced CR or PR as assessed by investigator is reported.
Time Frame: Up to approximately 24 months
Population: All participants who received at least 1 dose of study treatment. Per protocol, the 1 participant who switched over from Arm 1 Part 1: V941 Monotherapy to Arm 2 Part 1: V941 + Pembrolizumab was excluded from Arm 2 Part 1: V941 + Pembrolizumab for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 3 | 15 | 20 | 16 | 16
Percentage of Participants | 0.0 [0.0 to 70.8] | 6.7 [0.2 to 31.9] | 5.0 [0.1 to 24.9] | 12.5 [1.6 to 38.3] | 0.0 [0.0 to 20.6]

5. Secondary Outcome: Presence of Mutant Kirsten Rat Sarcoma (KRAS) Specific T Cells
Description: The presence of mutant KRAS specific T cells (G12D, G12V, G13D, G12C, and Wild type) in blood was assessed using an enzyme linked immunosorbent spot (ELISpot) assay. ELISpot detects interferon gamma (IFN-g) producing T-cells in a participant's peripheral blood mononuclear cells (PBMC) in response to KRAS specific stimulation. Data are presented as spot forming cells (SFC) per 10^6 PBMC. The post-treatment ELISpot readout for a cycle is reported. A cycle is 3 weeks.
Time Frame: Cycle 1 - Cycle 9 (a cycle is 3 weeks) and at the Discontinuation Visit (at the time of withdrawal or up to 30 weeks, whichever occurs first)
Population: Participants with centrally-confirmed tumor KRAS mutations, with a baseline scan that demonstrated measurable disease and who received at least 1 dose of study treatment. The number of participants analyzed indicates a pre-treatment ELISpot readout for a cycle and a post-treatment ELISpot readout for a cycle, which are required for a participant's data to be reported for a particular cycle. A cycle is 3 weeks.
Measure: Mean (Standard Deviation); unit: Log10(IFN-g (SFC per 10^6 PBMC))
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 2 | 11 | 6 | 7 | 3
Log10(IFN-g (SFC per 10^6 PBMC))
  KRAS G12D Cycle 1: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  KRAS G12D Cycle 1 | 1.00 (NA) — Standard deviation was not calculatable when n<2. | 0.56 (0.45) |  |  |
  KRAS G12D Cycle 2: number analyzed (Participants) | 1 | 6 | 0 | 0 | 0
  KRAS G12D Cycle 2 | 0.60 (NA) — Standard deviation was not calculatable when n<2. | 0.59 (0.49) |  |  |
  KRAS G12D Cycle 3: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  KRAS G12D Cycle 3 | 1.45 (NA) — Standard deviation was not calculatable when n<2. | 0.76 (0.28) |  |  |
  KRAS G12D Cycle 4: number analyzed (Participants) | 0 | 2 | 6 | 3 | 3
  KRAS G12D Cycle 4 |  | 1.35 (0.80) | 2.08 (0.48) | 1.70 (0.82) | 2.14 (0.82)
  KRAS G12D Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 2 | 2
  KRAS G12D Cycle 6 |  |  | 2.34 (0.40) | 2.30 (0.53) | 2.34 (0.15)
  KRAS G12D Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G12D Discontinuation Visit | 0.54 (0.34) |  |  |  |
  KRAS G12V Cycle 1: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  KRAS G12V Cycle 1 |  | 0.59 (0.53) |  |  |
  KRAS G12V Cycle 2: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  KRAS G12V Cycle 2 | 0.90 (NA) — Standard deviation was not calculatable when n<2. | 0.12 (0.27) |  |  |
  KRAS G12V Cycle 3: number analyzed (Participants) | 0 | 5 | 0 | 0 | 0
  KRAS G12V Cycle 3 |  | 0.88 (0.54) |  |  |
  KRAS G12V Cycle 4: number analyzed (Participants) | 0 | 3 | 5 | 3 | 1
  KRAS G12V Cycle 4 |  | 1.84 (0.14) | 2.04 (1.17) | 1.94 (0.67) | 2.25 (NA) — Standard deviation was not calculatable when n<2.
  KRAS G12V Cycle 6: number analyzed (Participants) | 0 | 0 | 3 | 2 | 0
  KRAS G12V Cycle 6 |  |  | 1.64 (1.43) | 1.77 (0.21) |
  KRAS G12V Cycle 7: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  KRAS G12V Cycle 7 |  | 2.20 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  KRAS G12V Cycle 9: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  KRAS G12V Cycle 9 |  | 2.20 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  KRAS G12V Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G12V Discontinuation Visit | 1.45 (0.04) |  |  |  |
  KRAS G12C Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  KRAS G12C Cycle 1 |  | 0.78 (0.67) |  |  |
  KRAS G12C Cycle 2: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  KRAS G12C Cycle 2 | 0.00 (NA) — Standard deviation was not calculatable when n<2. | 0.60 (0.85) |  |  |
  KRAS G12C Cycle 3: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  KRAS G12C Cycle 3 |  | 1.10 (0.70) |  |  |
  KRAS G12C Cycle 4: number analyzed (Participants) | 0 | 2 | 5 | 4 | 1
  KRAS G12C Cycle 4 |  | 1.93 (0.72) | 2.07 (1.18) | 2.12 (0.89) | 2.45 (NA) — Standard deviation was not calculatable when n<2.
  KRAS G12C Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 3 | 0
  KRAS G12C Cycle 6 |  |  | 1.93 (1.29) | 2.24 (0.68) |
  KRAS G12C Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G12C Discontinuation Visit | 1.55 (0.35) |  |  |  |
  KRAS G13D Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  KRAS G13D Cycle 1 |  | 0.65 (0.49) |  |  |
  KRAS G13D Cycle 2: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  KRAS G13D Cycle 2 | 0.00 (NA) — Standard deviation was not calculatable when n<2. | 0.62 (0.56) |  |  |
  KRAS G13D Cycle 3: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  KRAS G13D Cycle 3 |  | 0.91 (0.87) |  |  |
  KRAS G13D Cycle 4: number analyzed (Participants) | 0 | 2 | 5 | 3 | 1
  KRAS G13D Cycle 4 |  | 1.92 (0.71) | 1.53 (1.02) | 1.48 (0.20) | 1.26 (NA) — Standard deviation was not calculatable when n<2.
  KRAS G13D Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 2 | 0
  KRAS G13D Cycle 6 |  |  | 1.60 (1.12) | 1.75 (0.05) |
  KRAS G13D Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G13D Discontinuation Visit | 0.92 (0.87) |  |  |  |
  Wild Type Cycle 1: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  Wild Type Cycle 1 | 1.08 (NA) — Standard deviation was not calculatable when n<2. | 0.24 (0.54) |  |  |
  Wild Type Cycle 2: number analyzed (Participants) | 1 | 10 | 0 | 0 | 0
  Wild Type Cycle 2 | 0.00 (NA) — Standard deviation was not calculatable when n<2. | 0.49 (0.60) |  |  |
  Wild Type Cycle 3: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  Wild Type Cycle 3 | 1.15 (NA) — Standard deviation was not calculatable when n<2. | 0.86 (0.60) |  |  |
  Wild Type Cycle 4: number analyzed (Participants) | 0 | 3 | 6 | 7 | 3
  Wild Type Cycle 4 |  | 1.79 (0.59) | 1.64 (0.59) | 1.56 (0.47) | 1.26 (0.59)
  Wild Type Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 3 | 2
  Wild Type Cycle 6 |  |  | 1.38 (1.01) | 1.88 (0.24) | 1.59 (0.08)
  Wild Type Cycle 7: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Wild Type Cycle 7 |  | 2.33 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  Wild Type Cycle 9: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Wild Type Cycle 9 |  | 1.95 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  Wild Type Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Wild Type Discontinuation Visit | 0.80 (0.71) |  |  |  |

6. Secondary Outcome: Mean Change From Baseline in Quantity of Mutant KRAS Specific T Cells
Description: Mean change from baseline in the quantity of mutant KRAS specific T cells in blood was assessed using an enzyme linked immunosorbent spot (ELISpot) assay. ELISpot detects interferon gamma (IFN-g) producing T-cells in a participant's peripheral blood mononuclear cells (PBMC) in response to KRAS specific stimulation. Data are presented as spot forming cells (SFC) per 10^6 PBMC. The mean change is reported.
Time Frame: Baseline and Cycle 1 - Cycle 9 (a cycle is 3 weeks) and at the Discontinuation Visit (at the time of withdrawal or up to 30 weeks, whichever occurs first)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Log10(IFN-g (SFC per 10^6 PBMC))
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 2 | 11 | 6 | 7 | 3
Log10(IFN-g (SFC per 10^6 PBMC))
  KRAS G12D Cycle 1: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  KRAS G12D Cycle 1 | 1.00 (NA) — Standard deviation was not calculatable when n<2. | 0.46 (0.56) |  |  |
  KRAS G12D Cycle 2: number analyzed (Participants) | 1 | 6 | 0 | 0 | 0
  KRAS G12D Cycle 2 | 0.60 (NA) — Standard deviation was not calculatable when n<2. | 0.54 (0.48) |  |  |
  KRAS G12D Cycle 3: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  KRAS G12D Cycle 3 | 1.45 (NA) — Standard deviation was not calculatable when n<2. | 0.76 (0.28) |  |  |
  KRAS G12D Cycle 4: number analyzed (Participants) | 0 | 2 | 6 | 3 | 3
  KRAS G12D Cycle 4 |  | 1.35 (0.80) | 1.50 (0.56) | 0.94 (1.26) | 1.78 (1.44)
  KRAS G12D Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 2 | 2
  KRAS G12D Cycle 6 |  |  | 1.45 (0.67) | 1.61 (1.51) | 2.34 (0.15)
  KRAS G12D Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G12D Discontinuation Visit | -0.11 (0.58) |  |  |  |
  KRAS G12V Cycle 1: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  KRAS G12V Cycle 1 |  | 0.59 (0.53) |  |  |
  KRAS G12V Cycle 2: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  KRAS G12V Cycle 2 | 0.9 (NA) — Standard deviation was not calculatable when n<2. | 0.12 (0.27) |  |  |
  KRAS G12V Cycle 3: number analyzed (Participants) | 0 | 5 | 0 | 0 | 0
  KRAS G12V Cycle 3 |  | 0.88 (0.54) |  |  |
  KRAS G12V Cycle 4: number analyzed (Participants) | 0 | 3 | 5 | 3 | 1
  KRAS G12V Cycle 4 |  | 1.84 (0.14) | 2.04 (1.17) | 1.84 (0.71) | 2.25 (NA) — Standard deviation was not calculatable when n<2.
  KRAS G12V Cycle 6: number analyzed (Participants) | 0 | 0 | 3 | 2 | 0
  KRAS G12V Cycle 6 |  |  | 1.64 (1.43) | 1.62 (0.00) |
  KRAS G12V Cycle 7: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  KRAS G12V Cycle 7 |  | 2.20 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  KRAS G12V Cycle 9: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  KRAS G12V Cycle 9 |  | 2.20 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  KRAS G12V Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G12V Discontinuation Visit | 1.45 (0.04) |  |  |  |
  KRAS G12C Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  KRAS G12C Cycle 1 |  | 0.78 (0.67) |  |  |
  KRAS G12C Cycle 2: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  KRAS G12C Cycle 2 | 0.00 (NA) — Standard deviation was not calculatable when n<2. | 0.60 (0.85) |  |  |
  KRAS G12C Cycle 3: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  KRAS G12C Cycle 3 |  | 1.10 (0.70) |  |  |
  KRAS G12C Cycle 4: number analyzed (Participants) | 0 | 2 | 5 | 4 | 1
  KRAS G12C Cycle 4 |  | 1.93 (0.72) | 1.64 (1.26) | 1.68 (0.91) | 1.85 (NA) — Standard deviation was not calculatable when n<2.
  KRAS G12C Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 3 | 0
  KRAS G12C Cycle 6 |  |  | 1.10 (1.07) | 1.75 (0.95) |
  KRAS G12C Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G12C Discontinuation Visit | 1.55 (0.35) |  |  |  |
  KRAS G13D Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  KRAS G13D Cycle 1 |  | 0.26 (0.06) |  |  |
  KRAS G13D Cycle 2: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  KRAS G13D Cycle 2 | -0.3 (NA) — Standard deviation was not calculatable when n<2. | 0.62 (0.56) |  |  |
  KRAS G13D Cycle 3: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  KRAS G13D Cycle 3 |  | 0.41 (1.70) |  |  |
  KRAS G13D Cycle 4: number analyzed (Participants) | 0 | 2 | 5 | 3 | 1
  KRAS G13D Cycle 4 |  | 1.92 (0.71) | 1.28 (0.76) | 0.25 (0.22) | 1.26 (NA) — Standard deviation was not calculatable when n<2.
  KRAS G13D Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 2 | 0
  KRAS G13D Cycle 6 |  |  | 1.06 (0.73) | 0.55 (0.05) |
  KRAS G13D Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  KRAS G13D Discontinuation Visit | 0.77 (1.08) |  |  |  |
  Wild Type Cycle 1: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  Wild Type Cycle 1 | 1.08 (NA) — Standard deviation was not calculatable when n<2. | -0.23 (0.67) |  |  |
  Wild Type Cycle 2: number analyzed (Participants) | 1 | 10 | 0 | 0 | 0
  Wild Type Cycle 2 | 0.00 (NA) — Standard deviation was not calculatable when n<2. | 0.28 (0.59) |  |  |
  Wild Type Cycle 3: number analyzed (Participants) | 1 | 5 | 0 | 0 | 0
  Wild Type Cycle 3 | 1.15 (NA) — Standard deviation was not calculatable when n<2. | 0.45 (0.90) |  |  |
  Wild Type Cycle 4: number analyzed (Participants) | 0 | 3 | 6 | 7 | 3
  Wild Type Cycle 4 |  | 1.79 (0.59) | 1.32 (0.54) | 0.79 (0.90) | 0.76 (0.66)
  Wild Type Cycle 6: number analyzed (Participants) | 0 | 0 | 4 | 3 | 3
  Wild Type Cycle 6 |  |  | 0.90 (0.63) | 1.12 (0.54) | 0.99 (0.08)
  Wild Type Cycle 7: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Wild Type Cycle 7 |  | 2.33 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  Wild Type Cycle 9: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Wild Type Cycle 9 |  | 1.95 (NA) — Standard deviation was not calculatable when n<2. |  |  |
  Wild Type Discontinuation Visit: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Wild Type Discontinuation Visit | 0.80 (0.71) |  |  |  |

7. Other Pre Specified Outcome: T-cell Receptor (TCR) Clonality and Diversity
Description: TCR clonality and diversity in the periphery and tumor.
Time Frame: Up to approximately 24 months
Population: Data were not collected for this outcome measure.
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: All-cause mortality was reported on all enrolled participants. Non-serious and serious AEs were reported on all participants who received at least one dose of study treatment. MedDRA preferred terms "Neoplasm Progression", "Malignant Neoplasm Progression" and "Disease Progression" not related to the drug are excluded.
Groups:
- Part 1: V941 + Pembrolizumab (Switched Over From V941 Monotherapy): Participants who received the initial treatment of V941(mRNA-5671/V941) 1 mg administered IM Q3W for 9 3-week cycles and developed progressive disease were eligible to switch over to V941 1 mg administered IM Q3W for 9 3-week cycles and pembrolizumab 200 mg, IV for 35 3-week cycles.
Arm/Group | Part 1: V941 Monotherapy | Part 1: V941 + Pembrolizumab | Part 1: V941 + Pembrolizumab (Switched Over From V941 Monotherapy) | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 1/3 | 12/15 | 1/1 | 13/20 | 12/16 | 13/16
Serious Adverse Events (participants affected / at risk) | 1/3 | 6/15 | 0/1 | 5/20 | 7/16 | 9/16
Other Adverse Events (participants affected / at risk) | 3/3 | 15/15 | 0/1 | 20/20 | 16/16 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: V941 Monotherapy (N=3) | Part 1: V941 + Pembrolizumab (N=15) | Part 1: V941 + Pembrolizumab (Switched Over From V941 Monotherapy) (N=1) | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) (N=20) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) (N=16) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab) (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: V941 Monotherapy (N=3) | Part 1: V941 + Pembrolizumab (N=15) | Part 1: V941 + Pembrolizumab (Switched Over From V941 Monotherapy) (N=1) | Part 2: Expansion Cohort 1 Non-small Cell Lung Cancer (V941 + Pembrolizumab) (N=20) | Part 2: Expansion Cohort 2 Colorectal Cancer (V941 + Pembrolizumab) (N=16) | Part 2: Expansion Cohort 3 Pancreatic Adenocarcinoma (V941 + Pembrolizumab) (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 4 (4) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 6 (16) | 1 (1)
Fatigue (General disorders) | 2 (3) | 4 (4) | 0 (0) | 4 (4) | 3 (3) | 8 (8)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 3 (3) | 0 (0) | 13 (32) | 10 (22) | 8 (8)
Injection site reaction (General disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 4 (17) | 4 (5)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (6) | 0 (0) | 13 (24) | 10 (35) | 10 (11)
Vaccination site pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 3 (6) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 3 (6) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03948763/Prot_SAP_000.pdf